CLINICAL TRIAL: NCT00553007
Title: The Relation Between Periodontal Disease and Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aichi Gakuin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGU070001
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Periodontal Disease; Metabolic Syndrome
Keywords: Periodontal disease; Metabolic Syndrome
MeSH Terms: conditions — Periodontal Diseases; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Periodontal therapy — Normal periodontal therapy is performed.

SUMMARY:
Periodontal disease is associated with the components of Metabolic syndrome, such as obesity, diabetes, hypertension and hyperlipidemia. Therefore, strong relation with periodontal disease and metabolic syndrome is suggested. the overall goal of this study is to define the relation between periodontal disease and metabolic syndrome, including atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periodontal disease

Exclusion Criteria:

* Patients with malignant disease
* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
features of periodontal disease and metabolic syndrome | one year

SECONDARY OUTCOMES:
Pulse wave velocity; max Intima-Media Thickness(IMT); mean IMT; ankle-brachial blood pressure index; toe-brachial blood pressure index | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuaki Matsubara, MD. PhD, Principal Investigator — Aichi Gakuin University
Locations (1):
- Aichi Gakuin University, Nagoya, Aichi-ken, Japan